CLINICAL TRIAL: NCT02704910
Title: Lateral Postural Inclination in Parkinson's Disease : Involvement of the Basal Ganglia ?
Acronym: IPOLAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not more patient with lateral deviation
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1131; ID RCB (Registry Identifier: 2011-A01533-38)
Record Dates: First submitted 2012-02-20; First posted 2016-03-10 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voluntary subject (Placebo Comparator): Patient without parkinson disease, without deep brain stimulation
  Interventions: Behavioral: Subthalamic stimulation
- Patients (Active Comparator): Subthalamic stimulation
  Interventions: Behavioral: Subthalamic stimulation

INTERVENTIONS:
Behavioral: Subthalamic stimulation — Assess difference of amplitude (in degree) of the postural deviation between both condition of unilateral condition of subthalamic nucleus

SUMMARY:
The objective of this study is to assess the origins of lateral postural inclination presented by some Parkinson disease's patients.

Several mechanisms could cause lateral postural inclination. Available data allow to suggest three hypothesis: (troubles of tonus, perception of vertical perturbation, trouble of perception of corporal axis

DETAILED DESCRIPTION:
Inclusion Criteria:

* 30 to 75 years old patient
* Parkinson disease's diagnosed since 5 years
* Treated by deep brain stimulation
* Patient with at least 6 degree lateral deviation
* Without vestibular troubles nor peripheral sensorial trouble.

Exclusion Criteria:

* Dementia (Mattis < 130 ou MMS <24), or severe depressive episode according to DSM IV-R criteria
* Camptocormia or incompatible anteflexion with the dispositive of measure device
* Pregnant woman, nursing mother

ELIGIBILITY:
Inclusion Criteria:

* 30 to 75 years old patient
* Parkinson disease's diagnosed since 5 years
* Treated by deep brain stimulation
* Patient with at least 6 degree lateral deviation
* Without vestibular troubles nor peripheral sensorial trouble.

Exclusion Criteria:

* Dementia (Mattis < 130 ou MMS <24), or severe depressive episode according to DSM IV-R criteria
* Camptocormia or incompatible anteflexion with the dispositive of measure device
* Pregnant woman, nursing mother

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Lateropulsion measured by computerized Posturography | 4 days
  The postural inclination is measured in two conditions: With and without Deep Brain Stimulation. (Gissot et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krack, MD, Study Director — University Hospital, Grenoble
Locations (2):
- France (2):
  - CHU de Grenoble - Médecine Physique et de Réadapatation, Grenoble
  - CHU de Grenoble - Unité des troubles du mouvement, Grenoble